CLINICAL TRIAL: NCT00793806
Title: Immunologic Abnormalities, Chronic Inflammation and Oxidative Stress in Chronic Kidney Disease
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Collaborators: Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, Madeleine Pahl, M.D., Associate Professor of Medicine and Director of the Renal Clinic, University of California, Irvine
Other Study IDs: 20075572
Record Dates: First submitted 2008-11-14; First posted 2008-11-19 (Estimated); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Chronic Kidney Disease
Keywords: chronic kidney disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Medical Tool: Diffuse Optical Spectroscopy measurements will be compared to a variety of laboratory parameters routinely measured in Chronic Inflammation and Oxidative Stress in Chronic Kidney Disease
  Interventions: Device: Diffuse Optical Spectroscopy

INTERVENTIONS:
Device: Diffuse Optical Spectroscopy — Diffuse Optical Spectroscopy measurements will be compared to a variety of laboratory parameters routinely measured in Chronic Inflammation and Oxidative Stress in Chronic Kidney Disease
  Other Names: Diffuse Optical Spectroscopy measurements

SUMMARY:
The common causes of mortality are late stages of chronic kidney disease, cardiovascular disease and infections, are associated with abnormalities of the immune system, an underlying state of chronic inflammation and oxidative stress. These processes have not been carefully described in the chronic kidney disease population. The researcher can use Diffuse Optical Spectroscopy to determine the immune system in individuals with chronic kidney disease and describe the association with chronic inflammation and oxidative stress in that population.

DETAILED DESCRIPTION:
The Diffuse Optical Spectroscopy can measure the absolute concentrations of reduced and oxygenated hemoglobins,cardiac output, mean arterial pressure, blood loss,blood hemoglobin concentration, water and lipid concentrations of the tissue.

The researchers can use Diffuse Optical Spectroscopy to monitor volume changes during the hemodialysis treatment and to correlate the changes in volume and blood pressure with the measures of oxidative stress and inflammation used in this study. The researchers can use Diffuse Optical Spectroscopy data to compare to laboratory parameters routinely measured to clinical parameters such as cause of chronic kidney disease, blood pressure and dialysis-related parameters.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older with chronic kidney disease undergoing hemodialysis have been treated with hemodialysis for at least 3 months
* 18 years and older for control

Exclusion Criteria:

* acute kidney disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2008-08; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Medical Tool | 4 weeks
  Diffuse Optical Spectroscopy measure blood values changes during the hemodialysis treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Madeleine Pahl, M.D., Principal Investigator — University of California, Irvine
Locations (3):
- United States (3):
  - Beckman Laser Institute, Irvine, California
  - University of California Medical Center: Dialysis Unit, Orange, California
  - UCIMC Dialysis center, Orange, California